CLINICAL TRIAL: NCT06701864
Title: Palpation Versus Ultrasonography for Identifying the Cricothyroid Membrane of Distorted Neck-anatomy
Acronym: DEVITRACH3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Robin Lohse, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: F-22064259-3
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Airway Management; Identification of the Cricothyroid Membrane
Keywords: Airway Management; Ultrasound; Palpation; Cricothyroid membrane
MeSH Terms: interventions — Palpation; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Randomised to either "palpation" or "ultrasonography"
  The participants are thus randomised to use either "palpation" or to use "ultrasonography" to DIAGNOSE the position of the cricothyroid membrane
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palpation (Active Comparator): digital palpation used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: Palpation
- Ultrasound (Experimental): Ultrasonography (either "String of pearls" or TACA approach) used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Palpation — Identification of the cricothyroid membrane using PALPATION, a procedure used to prepare for front of neck airway access
  Arms: Palpation
Diagnostic Test: Ultrasound — Identification of the cricothyroid membrane, using ULTRASONOGRAPHY with either the "String of pearls" or TACA aproach as chosen by the participant , a procedure used to prepare for front of neck airway access
  Arms: Ultrasound

SUMMARY:
Participants will be anesthesiologists, who will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography.

The participants can choose either the "String of pearls" or Thyroid-Airline-Cricoid-Airline (TACA) for the ultrasonographic method to be used .

The silicone model of the neck is distorted with with the larynx deviated to one of the sides to simulate a patient with neck pathology.

DETAILED DESCRIPTION:
Participants will be anesthesiologists, who will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography.

The participants can choose either the "String of pearls" or Thyroid-Airline-Cricoid-Airline (TACA) for the ultrasonographic method to be used .

The silicone model of the neck is distorted with with the larynx deviated to one of the sides to simulate a patient with neck pathology.

The test persons are randomized to use other palpation or ultrasonography. All attempts are video-taped.

ELIGIBILITY:
Inclusion Criteria:

* Participants in a airway management course

Exclusion Criteria:

* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Correct identification of the cricothyroid membrane within a minute | Within 1 minute during procedure
  The fraction of correct identifications of the location of the cricothyroid membrane

SECONDARY OUTCOMES:
Correct identification of the sagittal plane within the airway | Within 1 minute during procedure
  The fraction of identifications that were within the sagittal boundaries of the trachea

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No